CLINICAL TRIAL: NCT03082430
Title: Study GO-PRP: Assessing the Efficacy of Intra Articular Injection of Platelets Rich Plasma for Gonarthrosis Treatment in Routine Care
Brief Title: GO PRP: Assessing the Efficacy of Intra Articular Injection of Platelets Rich Plasma for Gonarthrosis Treatment in Routine Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Principal Investigator, Denis Arniaud, MD, Hospital St. Joseph, Marseille, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO PRP
Record Dates: First submitted 2017-03-06; First posted 2017-03-17 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: descriptive study
Masking Description: study for knee osteoarthritis patients treated in the center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- knee osteoarthritis patients. (Other): therapeutic management of symptomatic knee osteoarthritis (resistant to medical first-line treatment) by intra-articular injection of autologous PRP prepared in the same procedure and using a dedicated CE marked medical device and a validated and reproducible method of preparation.
  Interventions: Biological: autologous PRP.

INTERVENTIONS:
Biological: autologous PRP. — one autologous PRP patient in this study and monitor and follow the evolution of pain and the knee function

SUMMARY:
This monocentric protocol is designed to evaluate the efficacy of therapeutic management of symptomatic knee osteoarthritis (resistant to medical first-line treatment) by intra-articular injection of autologous PRP prepared in the same procedure and using a dedicated CE marked medical device and a validated and reproducible method of preparation

DETAILED DESCRIPTION:
The main objective is to get a 50% proportion of responders defined by answers "absent" or "light" in the KOOS questionnaire on questions about pain and difficulty walking on flat ground.

Secondary objectives include the safety validation of the use of PRP (prepared standardized manner by means of a given medical device) as second-line standard of care for osteoarthritis by the introduction of a systematic monitoring; and the feasibility of the health care system dedicated to the treatment of knee osteoarthritis by autologous PRP.

Furthermore, the secondary objectives are to monitor and follow the evolution of pain (VAS) and the knee function (KOOS score) at 1 month, 3 months, 6 months. Evaluation of MRI will be performed within 15 days prior (inclusion visit) injection and 6 months to assess the cartilage thickness and visualize a regenerative effect.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 20 to 80 years
* Gonarthrosis diagnostic objectified by the criteria of the American College of Rheumatology
* Joint pain for more than 6 months
* Answer "moderate" to the question about pain walking on flat ground
* Answer "moderate" to the question about trouble walking on flat ground
* Osteoarthritis stage 2 or 3 on the scale of Kellgren Lawrence (objectified radiography) within 6 months previous inclusion
* Axial deformation of less than or equal to 5 ° lower limbs
* Informed consent signed by the patient
* HB> 10g / dl
* Beta-HCG negative at baseline
* Ability to perform the procedures in the follow-up (50 not walk on a flat surface and up / down stairs).
* Being affiliated to a system of health insurance

Exclusion criteria:

* Axial deformation > 5 °
* Ligamentous instability
* Significant injuries or target knee or knee surgery contralateral side in 12 months previous the inclusion visit
* Ligament reconstruction in the 12 months précédants the inclusion visit
* Need a cane or assistance to move
* BMI> 35
* Thrombocytopenia <150 G / L
* Thrombocytosis> 450 G / L
* Known thrombopathy
* Anemia HB <10g / dl
* Active infections to HIV 1 and 2, Agp24, HCV Ab, Ag and HbS AcHbc, Ac HTLV I and II, TPHA
* Chronic treatment with corticosteroids per os or older than 2 weeks
* Injection intra-articular corticosteroid of less than 2 months
* Intra-articular injection of hyaluronic acid of less than 6 months
* NSAIDs or antiplatelet agent of less than 15 days
* Inability to stop NSAIDs (including aspirin) 15 days before the injection and the week following the injection
* Fever or recent illness
* Autoimmune diseases
* Inflammatory arthritis
* Immune deficiency
* Infectious diseases
* Pregnant women
* Adults legally protected (under guardianship and trusteeship)
* People simultaneously participating in other biomedical research16. Inability

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-19 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
to monitor and follow the evolution of pain | prior,1 month, 3 months, 6 months
  VAS to monitor and follow the evolution of pain
to monitor and follow the evolution of the knee function | prior,1 month, 3 months, 6 months
  (KOOS score)
Evaluation of MRI | prior,1 month, 3 months, 6 months
  Evaluation will be performed within 15 days prior (inclusion visit) injection and 6 months to assess the cartilage thickness and visualize a regenerative effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint Joseph, Marseille, France

IPD SHARING:
Plan to Share IPD: No